CLINICAL TRIAL: NCT03677154
Title: A Phase I/II Trial of Mosunetuzumab (BTCT4465A) as Consolidation Therapy in Patients With Diffuse Large B-Cell Lymphoma Following First-Line Immunotherapy and as Monotherapy or in Combination With Polatuzumab Vedotin in Elderly/Unfit Patients With Previously Untreated Diffuse Large B-Cell Lymphoma
Brief Title: Trial of Mosunetuzumab (BTCT4465A) as Consolidation Therapy in Participants With Diffuse Large B-Cell Lymphoma Following First-Line Immunochemotherapy and as Monotherapy or in Combination With Polatuzumab Vedotin in Elderly/Unfit Participants With Previously Untreated Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO40554
Record Dates: First submitted 2018-09-11; First posted 2018-09-19 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Consolidation Therapy (Cohort A) (Experimental): Participants with a partial response to first-line chemotherapy will receive mosunetuzumab up to the recommended consolidation dose (RCD).
  Interventions: Drug: Mosunetuzumab Intravenous (IV); Drug: Tocilizumab
- Elderly/Unfit Previously Untreated Monotherapy (Cohort B) (Experimental): Elderly/unfit participants with previously untreated DLBCL will receive mosunetuzumab at the previously determined recommended phase II dose (RP2D).
  Interventions: Drug: Mosunetuzumab Intravenous (IV); Drug: Tocilizumab
- Elderly/Unfit Previously Untreated Combination Therapy (Cohort C) (Experimental): Elderly/unfit participants with previously untreated DLBCL will receive mosunetuzumab in combination with polatuzumab vedotin.
  Interventions: Drug: Mosunetuzumab Subcutaneous (SC); Drug: Polatuzumab Vedotin; Drug: Tocilizumab

INTERVENTIONS:
Drug: Mosunetuzumab Intravenous (IV) — Participants in cohorts A and B will receive IV mosunetuzumab.
  Arms: Consolidation Therapy (Cohort A); Elderly/Unfit Previously Untreated Monotherapy (Cohort B)
Drug: Mosunetuzumab Subcutaneous (SC) — Participants in Cohort C will receive SC mosunetuzumab.
  Arms: Elderly/Unfit Previously Untreated Combination Therapy (Cohort C)
Drug: Polatuzumab Vedotin — Participants in Cohort C will receive IV polatuzumab vedotin.
  Arms: Elderly/Unfit Previously Untreated Combination Therapy (Cohort C)
Drug: Tocilizumab — Participants will receive tocilizumab via IV as needed to manage severe cytokine release syndrome (CRS).

SUMMARY:
This study will evaluate the safety, pharmacokinetics, and preliminary efficacy of mosunetuzumab following first-line diffuse large B-cell lymphoma (DLBCL) immunochemotherapy in participants with a best response of stable disease or partial response, or in elderly/unfit participants with previously untreated DLBCL, or subcutaneous mosunetuzumab in combination with polatuzumab vedotin IV in elderly/unfit participants with previously untreated DLBCL.

ELIGIBILITY:
Inclusion Criteria for All Cohorts

* At least one bi-dimensionally measurable nodal lesion, defined as > 1.5 cm in its longest dimension, or one bi-dimensionally measurable extranodal lesion, defined as > 1.0 cm in its longest diameter
* Adequate hematologic function
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2; with the exception of South Korea, where participants 80 years or older with ECOG >/= 2 will not be eligible

Inclusion Criteria Specific to Cohort A

Participants in Cohort A must also meet the following criteria for study entry:

* Histologically confirmed DLBCL according to World Health Organization (WHO) 2016 expected to express the cluster of differentiation-20 (CD20) antigen
* One prior therapy with any systemic anthracycline-based chemoimmunotherapy containing regimen for previously untreated DLBCL
* Best response of SD or PR to prior systemic chemoimmunotherapy at the end of induction treatment in accordance with the Lugano 2014 criteria

Inclusion Criteria Specific to Cohorts B and C

Participants in Cohorts B and C must also meet the following criteria for study entry:

* Previously untreated, histologically confirmed, DLBCL according to WHO 2016 classification
* Age >/= 80 years, or
* Age 65-79 years and considered ineligible for chemoimmuotherapy (R-CHOP) with at least one of the following: Impairment in at least two activity of daily living (ADL) components as defined in the protocol; impairment in at least two instrumental ADL components as defined in the protocol; cumulative illness rating scale - geriactic (CIRS-G) score of at least one cormorbidity with a severity score of 3-4 (not including lymphoma and hematologic deficiencies due to lymphoma) or a score of 2 in >/= 8 comorbidities; impairment in cardiac function, renal function, liver function, or other comorbidities such that the participant is unfit for full-dose immunochemotherapy, such as rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP)
* Participants with an initial ECOG performance status of 3 may be considered during screening if the performance status is DLBCL-related and if pre-phase treatment during the screening phase (not more than 100 mg/day up to 7 days prior to Cycle 1 Day 1) results in an improvement of ECOG performance status to </= 2 prior to enrollment

Exclusion Criteria for All Cohorts

Participants who meet any of the following criteria will be excluded from study entry:

* Transformed lymphoma
* CNS lymphoma
* Prior treatment with mosunetuzumab
* Prior stem cell transplant (autologous and allogeneic)
* History of confirmed progressive multifocal leukoencephalopathy (PML)
* Known or suspected chronic active Epstein Barr virus (CAEBV), hepatitis B, hepatitis C (HCV), or Human Immunodeficiency Virus (HIV)
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* Positive SARS-CoV-2 antigen or PCR test within 30 days prior to Cycle 1 Day 1
* Prior solid organ transplantation
* Current or past history of central nervous system (CNS) disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Clinically significant history of liver disease
* Prior treatment with radiotherapy within 2 weeks prior to Cycle 1, Day 1 (C1D1)
* Significant cardiovascular disease

Exclusion Criteria Specific to Cohort A

Participants in Cohort A who meet the following criteria will be excluded from study entry:

- Prior anti-lymphoma treatment with chemotherapy, immunotherapy, or biologic therapy 4 weeks prior to C1D1

Exclusion Criterion Specific to Cohorts B and C

Participants in Cohorts B and C who meet the following criterion will be excluded from study entry:

- Prior treatment for DLBCL with chemotherapy, immunotherapy, and biologic therapy

Exclusion Criteria Specific to Cohort C

Participants in Cohort C who meet the following criteria will be excluded from study entry:

- Current Grade >1 peripheral neuropathy by clinical examination or demyelinating form of Charcot-Marie-Tooth disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | Baseline through approximately 90 days after last study treatment
Positron Emission Tomography-Computed Tomography (PET-CT) Complete Response (CR) Rate at Time of Primary Response Assessment (PRA) According to Lugano 2014 Response Criteria (Cohort A) | 6-8 weeks after Cycle 8 Day 1 or the final dose of study treatment (cycle = 21 days)
PET-CT Objective Response Rate (ORR) at PRA According to Lugano 2014 Response Criteria as Determined by the Investigator (Cohort B) | 6-8 weeks after Cycle 8 Day 1 or the final dose of study treatment (cycle = 21 days)
PET-CT ORR at PRA According to the Lugano 2014 Criteria as Determined by an Independent Review Committee (IRC) (Cohort C) | 6-8 weeks after Cycle 8 Day 1 or the final dose of study treatment (cycle = 21 days)

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of Mosunetuzumab IV | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Minimum Serum Concentration (Cmin) of Mosunetuzumab IV | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Area Under the Curve (AUC) of Mosunetuzumab IV | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Clearance (CL) of Mosunetuzumab IV | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Volume of Distribution at Steady State (Vss) of Mosunetuzumab IV | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Maximum Serum Concentration (Cmax) of Mosunetuzumab SC | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Time to Maximum Serum Concentration (Tmax) of Mosunetuzumab SC | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Minimum Serum Concentration (Cmin) of Mosunetuzumab SC | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Area Under the Curve (AUC) of Mosunetuzumab SC | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Clearance (CL) of Mosunetuzumab SC | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Volume of Distribution at Steady State (Vss) of Mosunetuzumab SC | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Maximum Serum Concentration (Cmax) of Polatuzumab Vedotin IV | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Minimum Serum Concentration (Cmin) of Polatuzumab Vedotin IV | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Area Under the Curve (AUC) of Polatuzumab Vedotin IV | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Clearance (CL) of Polatuzumab Vedotin IV | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Volume of Distribution at Steady State (Vss) of Polatuzumab Vedotin IV | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
End of Infusion Concentration (Ceoi) of Polatuzumab Vedotin IV | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Trough Concentration (Ctrough) of Polatuzumab Vedotin IV | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
PET-CT Rate According to the Lugano 2014 Criteria at PRA as Determined by the Investigator (Cohorts B and C) and IRC (Cohort C) | 6-8 weeks after Cycle 8 Day 1 or the final dose of study treatment (cycle = 21 days)
Objective Response Rate (ORR), Defined as the Proportion of Participants with a Complete Response (CR) or Partial Response (PR) at PRA as Determined by the Investigator (Cohorts A and C) | Baseline through 2 years after PRA (up to a total of approximately 2.5 years)
Best ORR (CR or PR at any time) During the Study Based on PET-CT and/or CT Scans as Determined by the Investigator (All Cohorts) and by IRC (Cohort C) | Baseline through 2 years after PRA (up to a total of approximately 2.5 years)
Duration of Response (DOR) as Determined by the Investigator (All Cohorts) and by IRC (Cohort C) | From the first occurrence of a documented objective response to disease progression, relapse, or death, whichever occurs first (up to approximately 2.5 years)
Duration of Confirmed Response (DOCR) as Determined by the Investigator (All Cohorts) and by IRC (Cohort C) | From the first occurrence of a documented CR to disease progression or relapse, or death from any cause, whichever occurs first (up to approximately 2.5 years)
Progression-Free Survival (PFS) as Determined by the Investigator (All Cohorts) and by IRC (Cohort C) | From the first study treatment to the first occurrence of disease progression, relapse, or death, whichever occurs first (up to approximately 2.5 years)
Overall Survival (OS) | From the first study treatment to death from any cause
Time to Deterioration in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Physical Functioning and Fatigue (Cohorts B and C) | From the first study treatment to the first occurrence of disease progression, relapse, initiation of new anti-lymphoma treatment, or death from any cause, whichever occurs first (up to approximately 2.5 years)
Time to Deterioration in European Organization for Research and Treatment of Cancer Item Library (EORTC-IL17) Physical Functioning (Cohorts B and C) | From the first study treatment to the first occurrence of disease progression, relapse, initiation of new anti-lymphoma treatment, or death from any cause, whichever occurs first (up to approximately 2.5 years)
Time to Deterioration in the Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) Subscale (Cohorts B and C) | From the first study treatment to the first occurrence of disease progression, relapse, initiation of new anti-lymphoma treatment, or death from any cause, whichever occurs first (up to approximately 2.5 years)
Proportion of Participants Achieving a Clinically Meaningful Improvement in Physical Functioning as Measured by EORTC QLQ-C30 (Cohorts B and C) | From the first study treatment to the first occurrence of disease progression, relapse, initiation of new anti-lymphoma treatment, or death from any cause, whichever occurs first (up to approximately 2.5 years)
Proportion of Participants Achieving a Clinically Meaningful Improvement in Physical Functioning as Measured by EORTC IL17 (Cohorts B and C) | From the first study treatment to the first occurrence of disease progression, relapse, initiation of new anti-lymphoma treatment, or death from any cause, whichever occurs first (up to approximately 2.5 years)
Anti-Drug Antibodies (ADAs) to Mosunetuzumab | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)
Anti-Drug Antibodies (ADAs) to Polatuzumab Vedotin (Cohort C) | At pre-defined intervals from Cycle 1 Day 1 through approximately 90 days after the last study treatment (cycle = 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (32):
- United States (8):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - University of California, Los Angeles (UCLA) - Hematology/Oncology Santa Monica, Santa Monica, California
  - Fort Wayne Medical Institute, Fort Wayne, Indiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Duke University, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
- Israel (7):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Carmel medical center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Ein-Karem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Sheba Medical Center, Ramat Gan
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - PRATIA MCM Kraków, Krakow
  - Centrum Onkologii Ziemi Lubelskiej im. ?w. Jana z Dukli, Lublin
  - Szpital Wojewodzki w Opolu, Opole
- South Korea (6):
  - Pusan National University Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Yeouido St. Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
- Spain (6):
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Universitario Vall d Hebron, Barcelona
  - Institut Catala d Oncologia Hospitalet, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing